CLINICAL TRIAL: NCT02725710
Title: Gabapentin as an Adjunct to Perioperative Pain Management Regimens for Uterine Aspiration: a Randomized Controlled Trial
Brief Title: Gabapentin as an Adjunct to Perioperative Pain Management Regimens for Uterine Aspiration
Acronym: GABA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00063872
Record Dates: First submitted 2016-03-02; First posted 2016-04-01 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Other Abortion; Spontaneous Abortion
Keywords: uterine aspiration
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Placebo (Active Comparator): Usual perioperative pain management protocol PLUS placebo orally 1-2 hour prior to procedure.
  Interventions: Drug: Placebo
- Group 2: Gabapentin (Active Comparator): Usual perioperative pain management protocol PLUS 600mg Gabapentin administered orally 1-2 hour prior to procedure.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 600mg Gabapentin administered orally 1-2 hours prior to procedure
  Other Names: Neurontin
  Arms: Group 2: Gabapentin
Drug: Placebo — Identical looking pill to the 600mg Gabapentin pill administered orally 1-2 hours prior to procedure
  Other Names: sugar pill
  Arms: Group 1: Placebo

SUMMARY:
This is a randomized controlled double-blind placebo-controlled trial evaluating the impact of gabapentin given preoperatively on perioperative pain scores for women receiving uterine aspiration between 6 and 14+6 weeks gestation. This study will be a trial included in a prospective meta-analysis evaluating the use of gabapentin on perioperative pain in the abortion setting.

ELIGIBILITY:
Inclusion Criteria:

* Women >=18 years-old
* Presenting for a surgical abortion
* No contraindication to outpatient abortion
* No contraindication to gabapentin
* Fluency in English and able to provide informed consent

Exclusion Criteria:

* Allergy, sensitivity or contraindication to gabapentin
* Severe renal disease
* Currently using gabapentin or pregalabin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Gray, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray BA, Hagey JM, Crabtree D, Wynn C, Weber JM, Pieper CF, Haddad LB. Gabapentin for Perioperative Pain Management for Uterine Aspiration: A Randomized Controlled Trial. Obstet Gynecol. 2019 Sep;134(3):611-619. doi: 10.1097/AOG.0000000000003398. PMID 31403587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited between August 2016 and June 2018.
Pre-assignment Details: One subject randomized to gabapentin withdrew from the procedure.
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Started | 48 | 47
Completed | 47 | 47
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo | Group 2: Gabapentin | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.3) | 31.7 (6.1) | 31.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 95
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 43 | 44 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 95
Baseline Pain [Median (Inter-Quartile Range); unit: units on a scale] — Measured using the 100-mm visual analog scale (VAS), where 0 means no pain and 100 means worst pain in my life.
  units on a scale | 3.3 [0.5 to 22.3] | 3.0 [0.0 to 9.0] | 3.0 [0.0 to 14.0]

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on 100-mm VAS (Visual Analog Scale) at 5 Minutes Post-procedure
Description: Score range of 0 to 100, where 0 means no pain and 100 means worst pain in my life.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
score on a scale | 35.7 (27.5) | 37.1 (30.4)
Statistical Analysis 1: Comparison: Group 1: Placebo vs Group 2: Gabapentin; Test type: Other; p = 0.56, Regression, Linear

2. Secondary Outcome: Pain Score on the 100-mm VAS
Description: Measured at baseline, 10 minutes post-procedure, and 30 minutes post-procedure. Score range of 0 to 100, where 0 means no pain and 100 means worst pain in my life.
Time Frame: Baseline (pre-operatively immediately prior to the procedure), 10 minutes, 30 minute
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
units on a scale
  Baseline | 3.3 [0.5 to 22.3] | 3.0 [0.0 to 9.0]
  10 minutes | 19.8 [7.5 to 42.5] | 20.0 [3.0 to 47.5]
  30 minutes | 12.6 [3.3 to 30.8] | 9.5 [1.0 to 31.5]

3. Secondary Outcome: Perioperative Nausea as Measured by 100-mm VAS
Description: Score range of 0 to 100, where 0 means no nausea and 100 means worst nausea in my life.
Time Frame: Baseline (pre-operatively immediately prior to the procedure), 10 minutes, 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
units on a scale
  Baseline | 3.0 [0.0 to 12.5] | 3.0 [0.0 to 20.0]
  10 minutes | 2.5 [0.0 to 14.0] | 1.0 [0.0 to 15.0]
  30 minutes | 2.3 [0.0 to 10.8] | 1.0 [0.0 to 18.0]

4. Secondary Outcome: Number of Subjects Experiencing Perioperative Vomiting
Time Frame: Baseline (pre-operatively immediately prior to the procedure), 10 minutes, 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
Participants
  Baseline | 1 | 0
  10 minutes | 1 | 2
  30 minutes | 1 | 5

5. Secondary Outcome: Perioperative Anxiety as Measured by the 100-mm VAS
Description: Score range of 0 to 100, where 0 means no anxiety and 100 means extremely anxious.
Time Frame: 5 minutes, 10 minutes, 30 minutes, discharge
Population: One subject in the placebo group did not have anxiety at discharge measured.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
units on a scale
  5 minutes | 24.5 [10.0 to 50.5] | 23.5 [6.0 to 49.5]
  10 minutes | 14.5 [3.8 to 43.5] | 11.0 [4.0 to 36.0]
  30 minutes | 13.3 [2.8 to 25.0] | 7.0 [2.5 to 27.5]
  Discharge: number analyzed (Participants) | 47 | 47
  Discharge | 10.5 [2.0 to 27.0] | 8.0 [3.0 to 23.0]

6. Secondary Outcome: Number of Subjects Using Pain Medications
Description: Pain medications included ibuprofen and oxycodone.
Time Frame: 24 hours post-operatively
Population: The number of subjects analyzed for "ibuprofen and oxycodone" and "oxycodone only" reflects the number of subjects that received a prescription for opiates.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
Participants
  No pain medication | 10 | 17
  Ibuprofen only | 23 | 23
  Ibuprofen and oxycodone: number analyzed (Participants) | 32 | 38
  Ibuprofen and oxycodone | 9 | 6
  Oxycodone only: number analyzed (Participants) | 32 | 38
  Oxycodone only | 6 | 1

7. Secondary Outcome: Number of Subjects Experiencing Side Effects
Description: Side effects noted are dizziness, ataxia, somnolence, asthenia, headache, and amblyopia.
Time Frame: 10 minutes post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 48 | 47
Participants
  Dizziness | 14 | 20
  Ataxia | 8 | 6
  Somnolence | 37 | 41
  Asthenia | 31 | 27
  Headache | 5 | 5
  Amblyopia | 3 | 3

8. Secondary Outcome: Pain (on a 5-point Scale)
Time Frame: Post-operative day 1
Population: Data not collected.
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Nausea (on a 5-point Scale)
Time Frame: Post-operative day 1
Population: Data not collected.
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Vomiting (on a 5-point Scale)
Time Frame: Post-operative day 1
Population: Data not collected.
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Side Effects (on a 5-point Scale)
Time Frame: Post-operative day 1
Population: Data not collected.
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: General Satisfaction With the Procedure (on a 5-point Scale)
Time Frame: Post-operative day 1
Population: Data not collected.
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 minutes post-procedure
Arm/Group | Group 1: Placebo | Group 2: Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 40/48 | 43/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Placebo (N=48) | Group 2: Gabapentin (N=47)
Dizziness (Nervous system disorders) | 14 | 20
Ataxia (Nervous system disorders) | 8 | 6
Somnolence (General disorders) | 37 | 41
Asthenia (Nervous system disorders) | 31 | 27
Headache (Nervous system disorders) | 5 | 5
Amblyopia (Eye disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT02725710/Prot_SAP_000.pdf